CLINICAL TRIAL: NCT04557930
Title: Hopewell Hospitalist: A Video Game Intervention to Increase Advance Care Planning Conversations by Hospitalists With Older Adults
Brief Title: EFFICACY: Hopewell Hospitalist: A Video Game Intervention to Increase Advance Care Planning by Hospitalists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Sound Physicians (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Amber Barnato, Director of the Dartmouth Institute for Health Policy and Clinical Practices, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00031186; P01AG019783 (NIH)
Record Dates: First submitted 2020-09-11; First posted 2020-09-22 (Actual); Results first posted 2023-02-28 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: Advance Care Planning
Keywords: advance care planning; physician performance; serious games; narrative engagement

STUDY DESIGN:
Intervention Model Description: A stepped wedge crossover trial randomizing physician participants at the group level (i.e., hospital). Each hospital group 'crossed over' from control to intervention at a randomized time point.
Who Masked: Outcomes Assessor
Masking Description: A hospital's treatment assignment was masked during analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Control (No Intervention): The control arm occurred prior to receipt of the video game intervention. Each hospital group 'crossed over' from control to intervention at a randomized time point based on their assignment to the 'step' of the trial.
- Video Game Intervention (Experimental): Each hospital group 'crossed over' from control to intervention at a randomized time point. Physicians working at these hospitals, who agreed to participate in the trial, received a study iPad and were asked to play the video game loaded on the iPad for a minimum of 2 hours.
  Interventions: Behavioral: Hopewell Hospitalist Video Game

INTERVENTIONS:
Behavioral: Hopewell Hospitalist Video Game — Hopewell Hospitalist is a customized theory-based adventure video game that uses narrative engagement to educate physician players on advance care planning to increase physicians' likelihood of engaging in and billing for ACP conversations.
  Arms: Video Game Intervention

SUMMARY:
Hopewell Hospitalist is a theory-based adventure video game designed to increase the likelihood that a physician will engage in an advance care planning (ACP) conversation with a patient over the age of 65. Drawing on the theory of narrative engagement, players assume the persona of a hospitalist and navigate a series of clinical encounters with seriously-ill patients over the age of 65. Players experience the consequences of having (or not having) ACP conversations in a timely fashion. The planned study is a pragmatic stepped-wedge crossover phase III trial testing the efficacy of Hopewell Hospitalist for increasing ACP rates measured by ACP billing frequency.

DETAILED DESCRIPTION:
Introduction: Fewer than half of all people in the U.S. have a documented advance care plan, such as an advance directive, despite their importance in ensuring high-quality care at the end-of-life. Hospitalization offers an opportunity for physicians to initiate advance care planning (ACP) conversations. Despite expert recommendations, hospital-based physicians (hospitalists) do not routinely engage in these conversations, reserving them for the critically ill.

The objective of this study is to test the effect of a novel behavioral intervention on the incidence of ACP conversations by hospitalists practicing at a stratified random sample of hospitals drawn from 220 US acute care hospitals staffed by a large, nationwide acute care physician practice with an ongoing ACP quality improvement initiative.

Methods and analysis: We developed Hopewell Hospitalist, a theory-based adventure video game, to modify physicians' attitudes towards ACP conversations, and to increase their motivation for engaging in them. Drawing on the theory of narrative engagement, players assume the persona of Andy Jordan, a hospitalist who accepts a new job in a small town. Through a series of clinical encounters with seriously-ill patients over the age of 65, players experience the consequences of having (or not having) ACP conversations in a timely fashion. The planned study is a pragmatic stepped-wedge crossover phase III trial, testing the efficacy of Hopewell Hospitalist for increasing ACP conversations. We will randomize 40 hospitals to the month (step) in which they receive the intervention. We aim to recruit 30 hospitalists from up to 8 hospitals each step to complete the intervention, playing Hopewell Hospitalist for at least 2 hours on an iPad pre-loaded with the game. The primary outcome is ACP billing for patients age 65 and older managed by participating hospitalists. We hypothesize that the intervention will increase ACP billing in the quarter after dissemination, and have 80% power to detect a 1% absolute increase and 99% power to detect a 3.5% absolute increase.

Ethics and dissemination: Dartmouth's Committee for the Protection of Human Subjects has approved the study protocol, which is registered on clinicaltrials.gov. We will disseminate the results through manuscripts and the trials website. Hopewell Hospitalist will be made available on the iOS Application Store for download, free of cost, at the conclusion of the trial.

ELIGIBILITY:
Hospital Inclusion Criteria:

* Value-based delivery model of care (Bundled Payment Care Initiative)
* Staffed by Sound Physicians for at least 2 quarters
* Advance care planning billing rate in prior quarter greater than 0 percent
* Employs a nurse liaison
* Hospitalist chief approval to approach hospitalists

Hospital Exclusion Criteria:

* Sound Physicians no longer staffing the hospital
* Not staffed by Sound Physicians for at least 2 quarters
* Advance care planning billing rate in prior quarter of 0 percent
* Does not employ a nurse liaison
* Hospitalist chief disapproval to approach hospitalists
* Hospitalist chief does not provide contact information for hospitalists
* Target number of hospitalists for the "step" has been met or exceeded

Hospitalist Inclusion Criteria:

* Employed by Sound for at least 2 quarters and staffing an eligible hospital for at least 1 quarter
* ACP billing rate in prior quarter greater than 0 percent or answers eligibility question affirming use of ACP billing codes
* Provides informed consent
* Name matches a name in the contact list for the sample; OR is verified by communication through an employer-based email address
* Receipt of a functional iPad within study step time frame

Hospitalist Exclusion Criteria:

* Not employed by Sound for at least 2 quarters and staffing an eligible hospital for at least 1 quarter
* ACP billing rate in prior quarter of 0 percent or answers eligibility question refusing use of ACP billing
* Does not provide informed consent
* Provides consent after the given deadline for consenting
* Name does not match a name in the contact list for the sample; OR cannot be verified by communication through an employer-based email address
* Receipt of a nonfunctional iPad within study step time frame
* If the number of participants who consent per site exceeds targets, then participants who are part-time employees will be preferentially excluded

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amber Barnato, MD, MPH, MS, Principal Investigator — Dartmouth-Hitchcock Medical Center and Geisel School of Medicine�; Deepika Mohan, MD, MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified participant data and supporting information with other researchers upon request to the PI.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Upon publication of the planned manuscripts. Data will be retained through February 2028.
Access Criteria: Data will require completion of a data use agreement with Dartmouth.

REFERENCES:
- [Background] Mohan D, MacMartin MA, Chelen JSC, Maezes CB, Barnato AE. Development of a theory-based video-game intervention to increase advance care planning conversations by healthcare providers. Implement Sci Commun. 2021 Oct 13;2(1):117. doi: 10.1186/s43058-021-00216-8. PMID 34645515
- [Background] Mohan D, O'Malley AJ, Chelen J, MacMartin M, Murphy M, Rudolph M, Barnato A. Videogame intervention to increase advance care planning conversations by hospitalists with older adults: study protocol for a stepped-wedge clinical trial. BMJ Open. 2021 Mar 22;11(3):e045084. doi: 10.1136/bmjopen-2020-045084. PMID 33753443
- [Derived] Mohan D, O'Malley AJ, Chelen J, MacMartin M, Murphy M, Rudolph M, Engel JA, Barnato AE. Using a Video Game Intervention to Increase Hospitalists' Advance Care Planning Conversations with Older Adults: a Stepped Wedge Randomized Clinical Trial. J Gen Intern Med. 2023 Nov;38(14):3224-3234. doi: 10.1007/s11606-023-08297-y. Epub 2023 Jul 10. PMID 37429972

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates: July 2020-May 2021 Types of location: acute care hospitals
Pre-assignment Details: There was a minimum three month (maximum 7-month) run-in period prior to the exposure of patients to the physicians enrolled in the intervention. We distinguish below between physician participants who enrolled in the trial, and patient participants who were treated by physicians in the trial. The latter group were unconsented.
Units Other Than Participants: Hospital
Groups:
- Step 1: First group of hospitals randomized to receive the intervention. Pre-intervention phase lasted from Months 0-3; post-intervention phase lasted from Months 4-11
- Step 2: Second group of hospitals randomized to receive the intervention. Pre-intervention phase lasted from Months 0-4; post-intervention phase lasted from Months 5-11
- Step 3: Third group of hospitals randomized to receive the intervention. Pre-intervention phase lasted from Months 0-5; post-intervention phase lasted from Months 6-11
- Step 4: Fourth group of hospitals randomized to receive the intervention. Pre-intervention phase lasted from Months 0-6; post-intervention phase lasted from Months 7-11
- Step 5: Fifth group of hospitals randomized to receive the intervention. Pre-intervention phase lasted from Months 0-7; post-intervention phase lasted from Months 8-11
Period: Pre-intervention
Arm/Group | Step 1 | Step 2 | Step 3 | Step 4 | Step 5
Started (Physician participants who agreed to enroll in the trial) | 39; 8 Hospital | 30; 7 Hospital | 25; 6 Hospital | 41; 7 Hospital | 28; 7 Hospital
Patient Participants Treated by Enrolled Physician Participants | 3203; 8 Hospital | 2677; 7 Hospital | 3303; 6 Hospital | 4976; 7 Hospital | 6615; 7 Hospital
Completed (Physician participants who completed study tasks) | 39; 8 Hospital | 30; 7 Hospital | 25; 6 Hospital | 41; 7 Hospital | 28; 7 Hospital
Not Completed | 0; 0 Hospital | 0; 0 Hospital | 0; 0 Hospital | 0; 0 Hospital | 0; 0 Hospital
Period: Post-intervention
Arm/Group | Step 1 | Step 2 | Step 3 | Step 4 | Step 5
Started | 39; 8 Hospital | 30; 7 Hospital | 25; 6 Hospital | 41; 7 Hospital | 28; 7 Hospital
Patient Participants Treated by Enrolled Physicians | 8076; 8 Hospital | 4691; 7 Hospital | 3706; 6 Hospital | 3949; 7 Hospital | 3030; 7 Hospital
Completed (We used an intention to treat analysis, so all physician participants enrolled in the trial were deemed to have 'completed' the intervention. There was loss to follow up in only 1 step (Step 2). Two physicians here did not complete all study tasks.) | 39; 8 Hospital | 30; 7 Hospital | 25; 6 Hospital | 41; 7 Hospital | 28; 7 Hospital
Not Completed | 0; 0 Hospital | 0; 0 Hospital | 0; 0 Hospital | 0; 0 Hospital | 0; 0 Hospital

BASELINE CHARACTERISTICS:
Population: physicians who enrolled in the trial
Groups:
- Intervention: The control arm occurs prior to receipt of the video game intervention. Each hospital group 'crosses over' from control to intervention at a randomized time point.
Arm/Group | Intervention
Number analyzed (Participants) | 163
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 108
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 154
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 75
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 52
  More than one race | 0
  Unknown or Not Reported | 21
Region of Enrollment [Number; unit: participants]
  United States | 163
Physician Experience in Years of Practice [Mean (Standard Deviation); unit: years] | 6.7 (5)
How frequently do you use the Advance Care Planning [ACP] billing codes [Count of Participants; unit: Participants]
  Always | 54
  Often | 74
  Sometimes | 28
  Rarely | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Advance Care Planning Bills
Description: Percentage of advance care planning bills submitted by physicians in the trial for patients over the age of 65 in the period before and after the roll-out of the video game intervention at their hospital. Advance care planning bills are defined as the presence/absence of ACP charges (Medicare billing codes 99497 or 99498) during a patient's hospitalization.
Time Frame: 11 months
Population: We analyzed outcomes for patients over 65 admitted for an acute illness, and treated by a trial participant in the pre- and post-intervention periods.
Measure: Count of Participants; unit: Participants
Groups:
- Pre-intervention: Patients treated by trial participants before the roll-out of the intervention at their hospital.
- Post-intervention: Patients treated by trial participants after the roll-out of the intervention at their hospital.
Arm/Group | Pre-intervention | Post-intervention
Number analyzed (Participants) | 20,774 | 23,461
Participants | 5,298 | 4,920
Statistical Analysis 1: Comparison: Pre-intervention vs Post-intervention; We tested the association between exposure to the intervention and the incidence of ACP billing in the pre- and post-intervention periods using a mixed effects logistic regression model, adjusting for time, patient and hospital covariates; Test type: Superiority; p = 0.41, Mixed Models Analysis; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.88 to 1.06]
Statistical Analysis 2: Comparison: Pre-intervention vs Post-intervention; Test type: Superiority — Sensitivity analysis of the association between the intervention and ACP billing, adjusted for time, patient characteristics, hospital characteristics, and the interaction between step of the trial and the intervention; p = 0.74, Mixed Models Analysis; Overall effect allowing effect heterogeneity across steps <0.001 Interaction effect <0.001; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.89 to 1.19] — Step 1 cohort
Statistical Analysis 3: Comparison: Pre-intervention vs Post-intervention; Sensitivity analysis of the association between the intervention and ACP billing, adjusted for time, patient characteristics, hospital characteristics, and the interaction between step of the trial and the intervention; Test type: Superiority; p = 0.09, Mixed Models Analysis; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.98 to 1.36]; Step 2 cohort
Statistical Analysis 4: Comparison: Pre-intervention vs Post-intervention; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.11, Mixed Models Analysis; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.97 to 1.33]; Step 3 cohort
Statistical Analysis 5: Comparison: Pre-intervention vs Post-intervention; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Odds Ratio (OR) = 0.66, 95% CI 2-sided [0.57 to 0.76] — Step 4 cohort
Statistical Analysis 6: Comparison: Pre-intervention vs Post-intervention; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.49, Mixed Models Analysis; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.89 to 1.19]; Step 5 cohort

2. Secondary Outcome: Percentage of Patients Who Died While in Hospital
Description: Number of patients who died in the pre-intervention and post-intervention period/total number of patients for both periods
Time Frame: 11 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Control | Video Game Intervention
Number analyzed (Participants) | 20,774 | 23461
Participants | 1625 | 1862

3. Secondary Outcome: Percentage of Patients Readmitted in 7 Days
Description: Number of patients readmitted within 7 days/Total number of patients treated in the pre-intervention and post-intervention periods
Time Frame: 11 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Control | Video Game Intervention
Number analyzed (Participants) | 20,774 | 23,461
Participants | 756 | 750

4. Secondary Outcome: Percentage of Patients Readmitted Within 30-days
Description: Number of patients readmitted within 30-days/Total number of patients in the pre-intervention and post-intervention periods
Time Frame: 11 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Control | Video Game Intervention
Number analyzed (Participants) | 20,774 | 23,461
Participants | 2,065 | 2,190

5. Secondary Outcome: Percentage of Patients Who Received Critical Care
Description: Number of patients who received critical care while admitted/total number of patients admitted in the pre-intervention and post-intervention periods
Time Frame: 11 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Control | Video Game Intervention
Number analyzed (Participants) | 20,774 | 23,461
Participants | 1,065 | 1,034

6. Secondary Outcome: Length of Stay
Description: Duration of hospitalization for patients treated in the pre-intervention and post-intervention periods
Time Frame: 11 months
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Usual Care Control | Video Game Intervention
Number analyzed (Participants) | 20,774 | 23,461
Days | 6.5 (5.3) | 6.4 (5.0)

ADVERSE EVENTS:
Time Frame: 11 months
Groups:
- Pre-intervention: The control arm occurs prior to receipt of the video game intervention.
- Post-Intervention: Physicians in the hospital group receive an iPad with the intervention pre-loaded, that they are asked to play for at least 2 hours.
  Hopewell Hospitalist Video Game: Hopewell Hospitalist is a customized theory-based adventure video game that uses narrative engagement to educate physician players on advance care planning to increase physicians' likelihood of engaging in and billing for ACP conversations.
Arm/Group | Pre-intervention | Post-Intervention
All-Cause Mortality (participants affected / at risk) | 0/163 | 0/163
Serious Adverse Events (participants affected / at risk) | 0/163 | 0/163
Other Adverse Events (participants affected / at risk) | 0/163 | 0/163

LIMITATIONS AND CAVEATS:
Heterogeneity of treatment effect across steps of the trial, suggesting the possibility of confounding secondary to the impact of COVID on hospital conditions.

Other limitations include: 1) generalizability of the results; 2) bias from non-random patterns of missingness in the data; 3) failure to systematically evaluate the fidelity and implementation of the intervention as planned due to COVID.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-03-17): https://cdn.clinicaltrials.gov/large-docs/30/NCT04557930/Prot_001.pdf
  • Statistical Analysis Plan (2021-11-11): https://cdn.clinicaltrials.gov/large-docs/30/NCT04557930/SAP_002.pdf
  • Informed Consent Form (2020-03-11): https://cdn.clinicaltrials.gov/large-docs/30/NCT04557930/ICF_003.pdf